CLINICAL TRIAL: NCT05006729
Title: RURAL Study Coordinating Center and Pulmonary Core
Brief Title: Risk Underlying Rural Areas Longitudinal Cohort Study (RURAL) Heart and Lung Study
Acronym: RURAL
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vasan Ramachandran, Dean School of Public Health, The University of Texas Health Science Center at San Antonio
Other Study IDs: H-42363; U01HL146382 (NIH); HSC20230132H (Other: UT Health San Antonio)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Rural Health; Pulmonary Disease; Heart Diseases
Keywords: Risk factors for heart disease; Risk factors for lung disease; Psychosocial factors; Familial factors; Economic factors; Mobile examination unit (MEU); Alabama; Kentucky; Louisiana; Mississippi
MeSH Terms: conditions — Lung Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens will be de-identified. All phenotype and genotype information associated with the biospecimens may be shared in accordance with the NHLBI Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC) data repository sharing policies, in which investigators may obtain de-identified and limited data sets via formal agreements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RURAL cohort study: A longitudinal research project in ten rural counties in Alabama, Kentucky, Louisiana, and Mississippi enrolling approximately 4,600 participants from these communities, examining several different aspects of their health, including heart and lung function.

SUMMARY:
The University of Texas Health Science Center at San Antonio (UTHSCSA) will serve as the site for the RURAL Study Coordinating Center, led by PI Vasan Ramachandran, MD.

The primary function of the Study Coordinating Center (SCC) is to serve as an administrative liaison between all of the RURAL study's cores. The SCC schedules, facilitates, and hosts, all RURAL meetings including preparation for Observational Study Monitoring Board (OSMB) meetings, and maintains direct communication with the study's program officers at NHLBI. The SCC monitors the overall progress of RURAL and keeps all RURAL cores abreast of study updates through meetings, emails, newsletters. It also maintains the official RURAL website and serves as an administrator for investigators seeking to collaborate with RURAL through the submission of Ancillary Studies. The SCC will have no direct interaction with any participants, nor will it have access to identifiable data.

DETAILED DESCRIPTION:
The Risk Underlying Rural Areas Longitudinal (RURAL) Cohort is a health research project that plans to enroll approximately 4,600 adults in ten rural counties throughout Alabama (AL), Kentucky (KY), Louisiana (LA), and Mississippi (MS). The ten specific counties are: Dallas County, AL; Wilcox County, AL; Boyle County, KY; Perry County, KY; Garrard County, KY; Breathitt County, KY; Assumption Parish, LA; Franklin Parish, LA; Oktibbeha County, MS; and Panola County, MS. The study will help to better understand health and disease in these rural areas. The information gathered in this study will help build future health programs to improve the health of local people in your community, which may promote healthier lives. Several different aspects of the participants' health will be examined including heart and lung function.

Broad goals of the RURAL Cohort Study include:

* Identifying the frequency of and risk factors for heart and lung diseases in the RURAL communities
* Identifying unique factors contributing to health disorders in these communities - including psychosocial, economic, and familial factors - and how they interact together
* Identifying potential solutions by examining differences between higher and lower risk rural counties

Findings from the RURAL study will inform health care providers, participants, researchers and the community regarding the frequency, burden, determinants, and prognosis of heart, lung, blood, and sleep diseases in the rural South, provide new knowledge that is critical for rural implementation science, and set the stage for collaborative opportunities for a wider community of scientists.

Participants in the RURAL Study will receive information on different areas of their health, including their heart and lungs.

Investigators will visit participants in their communities to complete a research exam about heart and lung health. Participants will attend an in-person exam at the RURAL study mobile exam vehicle. On the mobile exam unit participants will also receive a Fitbit [activity tracker] device and a RURAL cell phone app that will be used to collect information about their health and lifestyle.

Participants will receive results from their research exam, which they can also share with their doctor. The RURAL Study team will refer participants to a health center if there are immediate health concerns found during the research exam.

The RURAL Study follows all HIPAA rules and regulations, in addition to the NIH and institutional guidelines, for the protection of all research participants. No information from the study that could identify a participant will be publicly shared.

The RURAL study team will track participants' physical activity using the provided Fitbit device. The RURAL health team will also ask questions about overall health and lifestyle through the RURAL cell phone app. Participants will receive a kit to measure environmental and health factors in your home.

The visit in the mobile exam vehicle will take about 3 hours and will include:

* Vital signs including height and weight
* Blood draw
* Interviews and surveys asking about lifestyle and health history
* Tests related to heart, lung, and blood vessel health

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of specific counties in Alabama, Kentucky, Louisiana, and Mississippi
* Have resided in the specific county for the past two years and plan to reside at the residence for the next two years
* Speak English or Spanish

Exclusion Criteria:

* Currently incarcerated or institutionalized
* Currently in hospice care with a terminal illness and less than 6 month life expectancy
* Being actively treated for cancer

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Risk Underlying Rural Areas Longitudinal (RURAL) Cohort is a health research project in ten rural counties throughout Alabama, Kentucky, Louisiana, and Mississippi of residents 25-64 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Risk factors for lung disease in rural areas | 5 years
Risk factors for heart disease in rural areas | 5 years

SECONDARY OUTCOMES:
Pulmonary function | 5 years
Heart function | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vasan Ramachandran, MD, Study Director — University of Texas Health Science Center San Antonio; Suzanne Judd, PhD, Principal Investigator — University of Alabama at Birmingham; Paul Targonski, MD PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The RURAL (Risk Underlying Rural Areas Longitudinal) Cohort Study aims to address critical gaps in our knowledge of heart and lung disorders in rural counties in the southeastern US. — https://www.theruralstudy.org/